CLINICAL TRIAL: NCT07330466
Title: Does Spinal Cord Stimulation (SCS) Have an Effect Beyond Patients' Expectations? An Investigation of Treatment and Placebo Effects
Brief Title: Does Spinal Cord Stimulation Have an Effect Beyond Patients' Expectations? An Investigation of Treatment and Placebo Effects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Christina Emborg, Postdoc, University of Aarhus
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Spinal Cord Stimulation; 3165-00146B (Other Grant/Funding Number: Independent Research Fund Denmark)
Record Dates: First submitted 2025-09-19; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-09

CONDITIONS: Spinal Cord Stimulation
Keywords: Spinal Cord Stimulation; Chronic pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo condition (Placebo Comparator): The patient is incorrectly told that stimulation is on
  Interventions: Device: Stimulation OFF; Device: Told ON
- Total treatment (Active Comparator): The patient is correctly told that stimulation is on
  Interventions: Device: Stimulation ON; Device: Told ON
- Stimulation treatment (Other): The patient is incorrectly told that stimulation is off
  Interventions: Device: Stimulation ON; Device: Told OFF
- Control condition (Other): The patient is correctly told that stimulation is off
  Interventions: Device: Stimulation OFF; Device: Told OFF

INTERVENTIONS:
Device: Stimulation ON — Stimulator will be turned on
  Arms: Stimulation treatment; Total treatment
Device: Stimulation OFF — Stimulation is turned off
  Arms: Control condition; Placebo condition
Device: Told ON — Verbal suggestion that stimulation is on
  Arms: Placebo condition; Total treatment
Device: Told OFF — Verbal suggestion that stimulation is off
  Arms: Control condition; Stimulation treatment

SUMMARY:
The aim of the study is to evaluate treatment outcomes of Spinal Cord Stimulation. In the study each patient participates in four test sessions of 4-5 hours. Patients arrive for test days with their stimulation on. In each test session, baseline pain is first evaluated. Then, SCS is regulated (on/off) and patients evaluate their pain intensity immidiately and every 15 minutes during the test sessions. Patients are blinded to the treatment conditions during their participation in the study. At all times, patients can resume their usual treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients (>18 years of age) with SCS implanted to treat chronic pain.
* Patients who consent to participation and can cooperate in the study.
* Use of continuous paresthesia-free SCS for minimum 6 months prior to participation in the study.
* Pain score of 7 or less on a 0-10 scale in the most painful area treated with SCS, rated upon inclusion.
* Patients not receiving other neuromodulation treatment.
* Patients who have not undergone changes in their (pain relevant) medication during the last 30 days (pro necessitate medication allowed).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Patients' subjective pain intensity evaluated on a 0-10 Mechanical Visual Analogue Scale (M-VAS) | From enrollment to completion of four test sessions scheduled with a minimum interval of one week between each session.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark